CLINICAL TRIAL: NCT04042415
Title: Calorie Restriction as a Novel Therapeutic Tool to Manipulate Immunity and Improve Therapeutic Potential of First Line Drug Treatments During Relapsing Remitting Multiple Sclerosis
Brief Title: Calorie Restriction in Multiple Sclerosis
Acronym: Calorie-MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Principal Investigator, Giuseppe Matarese, Professor, Principal investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FISM 2018/S/5
Record Dates: First submitted 2019-07-17; First posted 2019-08-02 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Caloric Restriction
Keywords: Multiple Sclerosis; Immuno-metabolism; Calorie restriction; Treg cells; Inflammation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Inflammation | interventions — Caloric Restriction; Milk; Glutens

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Free diet controls (No Intervention): Patients on free diet
- Caloric restriction (Experimental): Patients will be treated with a mild caloric restriction (15-20% caloric restriction)
  Interventions: Other: Caloric restriction
- Caloric restriction without cow's milk and gluten (Experimental): Patients will be treated with a mild caloric restriction (15-20% caloric restriction) with exclusion of cow's milk, its derivatives and gluten
  Interventions: Other: Caloric restriction without cow's milk and gluten

INTERVENTIONS:
Other: Caloric restriction — Patients will be treated with a diet regimen of mild caloric restriction (15-20% caloric restriction)
  Arms: Caloric restriction
Other: Caloric restriction without cow's milk and gluten — Patients will be treated with mild caloric restriction (15-20% caloric restriction) plus excluding from diet cow's milk, its derivatives and gluten.
  Arms: Caloric restriction without cow's milk and gluten

SUMMARY:
There is a strong relationship between metabolic state and immune tolerance through a direct control exerted on immune cells by specific intracellular nutrient-energy sensors. An increased "metabolic work load" represents a novel issue linking metabolism with loss of self-immune tolerance. Several disease-modifying drugs have been approved for Relapsing-remitting Multiple Sclerosis (RR-MS) treatments and have shown to reduce relapse rates by modulating immune responses; however, their impact on long-term disease progression and accrual of irreversible neurological disability remains largely unclear, underlining the need for novel therapeutic strategies. In this context, both acute fasting (AF) and chronic caloric restriction (CR) have been shown to improve experimental autoimmune encephalomyelitis (EAE). Despite this evidence, no specific studies have been performed to dissect at the cellular level the mechanism of action of CR in the context of autoimmunity and MS. This study aims at investigating this specific point in order to pave the way for a wider utilization of a nutritional approach to alter MS progression and activity. The aim of this study is to improve the outcome of RR-MS and the efficacy of first line drug treatments (ie. Copaxone or Tecfidera) by altering the metabolic state of the host via calorie restriction with the aim to re-equilibrate immune/inflammatory responses of patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune disorder characterized by central nervous system (CNS) inflammation, demyelination, and axonal damage. Its pathogenesis consists of an initial T cell priming against myelin antigens in secondary lymphoid organs (induction phase) followed by migration of auto-reactive T cells and other immune system cells through the blood brain barrier into the CNS (effector phase). MS attacks are self-limiting, illustrating the existence of a regulatory network in which regulatory T cells (Treg) play a key role. Treg cells, which comprise 5%-10% of peripheral cluster of differentiation (CD)4+ T cells, inhibit effector T cell responses and can suppress MS. One of the immune abnormalities observed in MS is a reduction in the number and suppressive functions of Tregs. Furthermore, an abnormal Treg proliferation and metabolic profile was described in MS patients characterized by altered interleukin (IL) 2- IL 2 receptor - STAT5 signaling, and activation of the mammilian target of rapamycin (mTOR) metabolic pathway. More recently, the risk of MS has been associated with several environmental factors, including obesity and diet. Current treatments are only partially effective in controlling disease activity in relapsing-remitting (RR)-MS patients and no drugs are available that prevent or slow the progressive forms of MS. There remains an urgent need for new and safe therapies for patients that do not respond optimally to current drug treatments. In recent times, it has become evident that the control of orexigenic and anorexigenic circuits not only affects the regulation of body weight but also dramatically influences other important physiological and dominant functions, including immune homeostasis. In particular, several cytokines, hormones, neuropeptides and transcription factors play relevant roles in both metabolism and immunity.

It has been shown that dietary intervention can alter autoimmune disease progression, indeed dietary indoles suppress delayed-type hypersensitivity by inducing a switch from pro-inflammatory Th17 cells to anti-inflammatory Treg cells. Recent reports have shown that caloric restriction (CR) can significantly increase the survival and reduce clinical progression in EAE. CR induces multiple metabolic and physiologic modifications, including anti-inflammatory, antioxidant, and neuroprotective effects that could be beneficial in MS. A recent report has shown that dietary restriction improves repopulation but impairs lymphoid differentiation capacity of hematopoietic stem cells in early aging, by inhibiting the proliferation of lymphoid progenitors, resulting in decreased production of peripheral B lymphocytes and impaired immune function. Moreover prolonged fasting (PF) or a fasting mimicking diet (FMD) lasting 2 or more days have been shown to increase protection of multiple systems against a wide variety of chemotherapy drugs; PF or FMD reverses the immunosuppression or immunosenescence effects of either chemotherapy or aging by a hematopoietic stem cell-based regenerative process. Chronic CR, a ketogenic diet (KD) and intermittent fasting have been shown to prevent EAE, reducing inflammation, demyelination, and axon injury - without suppressing immune functions, when administered prior to disease induction or signs. CR associates with increased plasma levels of corticosterone and adiponectin, and with reduced concentrations of IL-6 and leptin. The effects of CR in EAE in the monophasic Lewis rat model show that upon calories restriction by 33% or 66%, EAE can be totally inhibited in the latter group, in which a depressed immune function with fewer T cells in lymphoid organs, impaired proliferation and cytokine production are observed. CR could benefit EAE through multiple metabolic and cytokine/adipokine changes that ultimately lead to a reduced inflammatory response. Other possibilities include CR-associated increase in ghrelin, neuropeptide Y (NPY) and endocannabinoids - all of which can dampen EAE and are increased during CR and starvation. Environmental factors are believed to play a role in the pathogenesis of MS, which is more prevalent in the Western world, where increased intake of saturated fats of animal origin is common. Although there has been speculation that diet may alter the course of MS, only a few randomized, controlled studies of dietary alterations in autoimmunity have been published, and none involving CR. Yet, dietary intervention might be attractive in MS, i.e. with CR associated with adequate nutrition, which can be safely accomplished through proper monitoring and could provide additional benefits such as improved insulin sensitivity, lower low-density lipoprotein, cholesterol, blood pressure and, importantly, reduced inflammation.

In conclusion, in spite of the above robust experimental evidence, no specific studies have been performed to dissect at cellular level the mechanism of action of CR in the context of autoimmunity and MS. This study aims at investigating this specific point to pave for a wider utilization of the nutritional approach to alter MS progression and activity to be associated to first line drug treatments.

Rationale and specific aims.

Several disease modifying drugs are approved for RR-MS treatments and have shown to reduce relapse rates by modulating immune responses; however, their impact on long-term disease progression and accrual of irreversible neurological disability remains largely unclear, underlining the need for novel therapeutic strategies.

The aim of this pilot study is to investigate the cellular and molecular mechanism of action of metabolic manipulation through CR accompanied or not to removal of specific antigenic foods (gluten/cow's milk) and their impact on RR-MS progression during treatment with conventional first line drugs.

the objective of this study is to improve the outcome of RR-MS and the efficacy of first line drug treatments (either dimethyl fumarate or glatiramer acetate) by altering the metabolic state of the host via a mild CR (15-20% caloric restriction of the ideal diet for the individual) accompanied or not to removal of specific foods from diet (gluten and cow's milk derivatives), with the aim to re-equilibrate immune/inflammatory responses of the patients.

Specifically, will be analyzed the following read outs in patients before and after specific treatments:

Aim 1) The impact of CR on the immunophenotype of different subclasses of circulating immune cells from the blood of RR-MS patients, and its correlation with the clinical status of the patients (ie. disease duration, number of relapses since onset, grade of disability and severity based on expanded disability status score (EDSS), MS severity score (MSSS) as well as presence of disease activity based on MRI imaging (gadolinium enhancing lesions) and overall lesion burden (T2 lesion volume)), and immuno-metabolic parameters (ie. circulating leptin, adiponectin, adipokines, etc);

Aim 2) The capacity of CR to affect T cell and regulatory T cell function/activity (activation, proliferation, suppression, Foxp3 induction) and molecular signalling pathway involved and possibly altered upon T-cell receptor (TCR) stimulation (ERK-mTOR-p27kip1 etc);

Aim 3) The effect of CR on the metabolic asset of circulating T cell populations (ie. measurement of glycolysis, oxidative phosphorylation and fatty acid oxidation);

Aim 4) The advanced proteomic profile, including protein modifications such as phosphorylation, acetylation, methylation, ubiquitination and glycosylation in conventional T cells and Treg cells from RR-MS subjects;

Aim 5) The effect of CR on the composition of the intestinal microbiota in RR-MS patients.

Patients will be enrolled at diagnosis before starting "first line" drug treatment (either Tecfidera or Copaxone). After starting pharmacological treatments, patients will be randomized in the following 3 groups:

1. 40 naive to treatment RR-MS (30 on Tecfidera + 10 Copaxone treatment) Free Diet Controls (FD);
2. 40 naive to treatment RR-MS (30 on Tecfidera + 10 Copaxone treatment) on mild Caloric Restriction (15-20% caloric restriction);
3. 40 naive to treatment RR-MS (30 Tecfidera + 10 Copaxone treatment) on mild Caloric Restriction as above in which Cow's Milk and its derivatives and Gluten have been removed (15-20% caloric restriction- plus excluding from diet cow's milk, its derivatives and gluten).

The patients will be enrolled in 10-12 months and followed for 24 months. Each group will have an equal distribution in age, gender and body mass index. Blood samples for the cellular, molecular and metabolic assessment of immune cells as well as the flow-cytometric extended analyses and proteomics will be obtained at baseline (T0), months 6 (T1), months 12 (T2) and months 24 (T3) after baseline. Besides the immunological studies, blood aliquots will be used for routine blood tests to control for concomitant infections. For the same purpose, urinalysis will be obtained at each time point. MRI scans will be performed for clinical practice at screening (Visit 0) and at months 6 (Visit 2), months 12 (Visit 3) and months 24 (Visits 4).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with early diagnosis (no more than 2 years) of RR-MS according to the revised McDonald (2017) criteria;
* Subjects naïve-to-treatment;
* Subjects with EDSS between 0-5.5;
* No use of oral or systemic corticosteroids or adrenocorticotropic hormone (ACTH) within 30 days prior to screening visit;
* Subjects with BMI > 22 kg/m2 and BMI < 28 kg/m2;
* Willing to collect a food diary for one week and to donate a blood and stool samples;
* No antibiotic treatment within 3 months of enrolment;
* No immunosuppressive therapy;
* Signed informed consent.

Exclusion Criteria:

* Pregnancy and breast-feeding;
* History of alcohol or drug abuse;
* Serious psychiatric disorders;
* Any major medical problem that in the opinion of the investigator could bias the results (e.g. HIV infection) or affect adherence to the protocol;
* Subjects with inadequate haematological function (defined by leukocyte ≤ 2,0 x 109; platelets <100 x 109; haemoglobin <12 g/dl for female and <13 g/dl for male), liver function (defined by aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase > 2.0 times upper limit of normal), thyroid function (according to physician's discretion);
* Known hypersensitivity to gadolinium;
* Any other condition that would prevent the subject from undergoing a contrast-enhanced MRI scan;
* Any contra-indication according to the specific first line treatment for MS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change of the "no evident disease activity" (NEDA) from baseline clinical status of MS patients at 6, 12, and 24 months | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Evaluation of the "no evident disease activity" (NEDA) defined thanks to the evaluation of three components: (i) absence of confirmed disability progression (CDP), (ii) absence of relapses and (iii) absence of radiological activity before and after starting caloric restricted diet.

SECONDARY OUTCOMES:
Percentage of different immune cells populations (circulating immune cells, regulatory T cells, conventional T cells, etc.) | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Evaluation of the percentage of different subclasses of circulating immune cells in the blood of patients
Mitotic cell divisions of conventional T cells | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Evaluation of the amount of conventional T cell divisions in the presence or absence of regulatory T cells through evaluation of 3H-thymidine incorporation into new strands of chromosomal DNA
Glycolytic metabolism of T cells (mpH/min) | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Evaluation of Glycolysis (mpH/min) through measurement of Extracellular Acidification Rate (ECAR) of circulating T cell populations
Oxidative metabolism of T cells (pMol/min) | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Evaluation of oxidative phosphorylation (pMol/min) through measurement of Oxygen Consumption Rate (OCR) of circulating T cell populations
Circulating adipokines (pg/ml) | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Evaluation of the serum/plasma concentration (pg/ml) of circulating adipokines (Leptin, adiponectin, etc...)
Change in the expression level of molecules involved in the signalling pathway of T-cell receptor (TCR) | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Analysis of molecules involved in the signalling pathway after T-cell receptor (TCR) stimulation (ERK-mTOR-p27kip1 etc);
Change in the composition of the gut microbiota | T0: before intervention, T1: after 6 months of intervention, T2: after 12 months of intervention, T3: after 24 months of intervention
  Evaluation of the components of the gut microbiota before and after starting caloric restricted diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromed - Istituto Neurologico Mediterraneo Pozzilli, Pozzilli, IS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Rosa V, La Cava A, Matarese G. Metabolic pressure and the breach of immunological self-tolerance. Nat Immunol. 2017 Oct 18;18(11):1190-1196. doi: 10.1038/ni.3851. PMID 29044230
- [Result] Sanna V, Di Giacomo A, La Cava A, Lechler RI, Fontana S, Zappacosta S, Matarese G. Leptin surge precedes onset of autoimmune encephalomyelitis and correlates with development of pathogenic T cell responses. J Clin Invest. 2003 Jan;111(2):241-50. doi: 10.1172/JCI16721. PMID 12531880
- [Result] Matarese G, Carrieri PB, La Cava A, Perna F, Sanna V, De Rosa V, Aufiero D, Fontana S, Zappacosta S. Leptin increase in multiple sclerosis associates with reduced number of CD4(+)CD25+ regulatory T cells. Proc Natl Acad Sci U S A. 2005 Apr 5;102(14):5150-5. doi: 10.1073/pnas.0408995102. Epub 2005 Mar 23. PMID 15788534
- [Result] De Rosa V, Procaccini C, La Cava A, Chieffi P, Nicoletti GF, Fontana S, Zappacosta S, Matarese G. Leptin neutralization interferes with pathogenic T cell autoreactivity in autoimmune encephalomyelitis. J Clin Invest. 2006 Feb;116(2):447-55. doi: 10.1172/JCI26523. Epub 2006 Jan 12. PMID 16410832
- See also: Laboratory site — http://www.matareselab.it
- See also: Italian MS Foundation official site with reference of the Calorie-MS study — https://www.aism.it/alimentazione_tagliare_le_calorie_rallentare_la_sclerosi_multipla